CLINICAL TRIAL: NCT02068729
Title: A Comparison of Complication Rates Between Lateral Approaches to the Lumbar Spine: K2M RAVINE® Far Lateral System Versus NuVasive XLIF®
Brief Title: Comparison of Complication Rates Between Lateral Approaches to the Lumbar Spine
Acronym: RAVINE
Status: Terminated | Type: Observational
Why Stopped: The study was terminated early due to slow enrollment and difficulties with long-term follow-up
Sponsor: K2M, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CA-002
Record Dates: First submitted 2014-02-11; First posted 2014-02-21 (Estimated); Results first posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Degenerative Disc Disease; Grade 1 Spondylolisthesis
Keywords: degenerative disc disease; DDD; Grade 1 spondylolisthesis; spondylolisthesis; L2-S1
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
An evaluation of the incidence of complications resulting from far lateral spine surgery utilizing the K2M RAVINE® Lateral Access System (RAVINE) with ALEUTIAN® Lateral Interbody Spacer System versus literature reported results for the NuVasive XLIF® system (XLIF) in the treatment of degenerative disc disease (DDD) with up to Grade 1 spondylolisthesis.

DETAILED DESCRIPTION:
An evaluation of the incidence of complications resulting from far lateral spine surgery utilizing the K2M RAVINE® Lateral Access System (RAVINE) with ALEUTIAN® Lateral Interbody Spacer System versus literature reported results for the NuVasive XLIF® system (XLIF) in the treatment of degenerative disc disease (DDD) with up to Grade 1 spondylolisthesis at L2-S1 requiring surgical intervention at one or two contiguous levels. Safety will be assessed by the following: 1.) Evaluation of all adverse events including device related, procedure related and additional serious adverse events; 2.) Additional surgical intervention at the operative site including the need for removals, revisions, re-operations or supplemental fixation required to modify the device; and 3.) The incidence and severity of any psoas muscle injury, genital femoral nerve injury and lumbar plexus injury will be determined for all patients. Supplemental fixation of any kind may be included as long as the procedure is completed via a minimally invasive approach.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DDD with up to Grade 1 spondylolisthesis, confirmed clinically and radiographically, requiring surgical intervention at one or two contiguous levels between L2-S1
* Inadequate response to conservative medical care over a period of at least 6 months
* Willing and able to comply with the requirements of the protocol including follow-up requirements
* Willing and able to sign a study specific informed consent
* Skeletally mature and ≥ 18 years of age at the time of enrollment

Exclusion Criteria:

* Previous anterior/posterior/lateral spine surgery at the index level
* Previous posterior/lateral spine surgery (e.g., posterior element decompression) that destabilizes the lumbar spine
* Active systemic infection or infection at the operative site
* Co-morbid medical conditions of the spine or upper/lower extremities that may affect the lumbar spine neurological and/or pain assessment
* Metabolic bone disease such as osteoporosis that contradicts spinal surgery
* History of an osteoporotic fracture
* History of an endocrine or metabolic disorder (e.g., Paget's disease) known to affect bone and mineral metabolism
* Taking medications that may interfere with bony/soft tissue healing including chronic steroid use
* Known allergy to titanium, cobalt chrome or PEEK
* Rheumatoid arthritis or other autoimmune disease or a systemic disorder such as HIV, active hepatitis B or C or fibromyalgia
* Current medical condition (e.g., unstable cardiac disease, cancer) that may result in patient death or have an effect on outcomes prior to study completion
* Pregnant, or intend to become pregnant, during the course of the study
* Severe obesity (Body Mass Index > 40)
* Physical or mental condition (e.g., psychiatric disorder, senile dementia, Alzheimer's disease, alcohol or drug addiction) that would interfere with patient self-assessment of function, pain or quality of life
* Involved in current or pending spinal litigation where permanent disability benefits are being sought
* Incarcerated at the time of study enrollment
* Current participation in an investigational study that may impact study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for study enrollment will have a primary diagnoses limited to degenerative disc disease (DDD) with up to Grade 1 spondylolisthesis at L2-S1 requiring surgical intervention at one or two contiguous levels. Qualified patients will have confirmed failure of conservative therapy as well as plain film imaging studies. Subjects must be ≥ 18 years old at the time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2014-06; Primary Completion 2019-09-11 (Actual); Study Completion 2020-02-28 (Actual)

REFERENCES:
- [Background] Malham GM, Ellis NJ, Parker RM, Seex KA. Clinical outcome and fusion rates after the first 30 extreme lateral interbody fusions. ScientificWorldJournal. 2012;2012:246989. doi: 10.1100/2012/246989. Epub 2012 Nov 1. PMID 23213282
- [Background] Caputo AM, Michael KW, Chapman TM Jr, Massey GM, Howes CR, Isaacs RE, Brown CR. Clinical outcomes of extreme lateral interbody fusion in the treatment of adult degenerative scoliosis. ScientificWorldJournal. 2012;2012:680643. doi: 10.1100/2012/680643. Epub 2012 Sep 24. PMID 23049476
- [Background] Youssef JA, McAfee PC, Patty CA, Raley E, DeBauche S, Shucosky E, Chotikul L. Minimally invasive surgery: lateral approach interbody fusion: results and review. Spine (Phila Pa 1976). 2010 Dec 15;35(26 Suppl):S302-11. doi: 10.1097/BRS.0b013e3182023438. PMID 21160394
- [Background] Berjano P, Balsano M, Buric J, Petruzzi M, Lamartina C. Direct lateral access lumbar and thoracolumbar fusion: preliminary results. Eur Spine J. 2012 May;21 Suppl 1(Suppl 1):S37-42. doi: 10.1007/s00586-012-2217-z. Epub 2012 Mar 9. PMID 22402840

RESULTS

PARTICIPANT FLOW:
Groups:
- K2M RAVINE Lateral Access System: This treatment group included patients treated with the RAVINE system that had:
  1. A diagnosis of degenerative disc disease (DDD) with up to Grade 1 spondylolisthesis at L2-S1, confirmed clinically and radiographically, required surgical intervention.
  2. One or two contiguous levels that required surgical intervention.
  3. Inadequately responded to conservative medical care over a period of at least 6 months.
  4. An age at time of enrollment greater or equal to 18 years old.
Period: Overall Study
Arm/Group | K2M RAVINE Lateral Access System
Started | 131
Completed | 56
Not Completed | 75

BASELINE CHARACTERISTICS:
Groups:
- Demographics and Baseline Characteristics: This is a demographic and baseline characteristics of the patient population. This includes parameters such as Age, Gender, Height, Weight Body Mass Index (BMI) and Tobacco Usage.
Arm/Group | Demographics and Baseline Characteristics
Number analyzed (Participants) | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 77
  >=65 years | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 47
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The study Case Report Forms did not include Race/Ethnicity
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 125
Body Mass Index (BMI) [Mean (Standard Deviation); unit: lbs/(in^2)*703] | 28.48 (4.4)
Height [Mean (Standard Deviation); unit: inches] | 65.96 (3.9)
Weight [Mean (Standard Deviation); unit: pounds] | 177.2 (36.7)
Tobacco Use [Count of Participants; unit: Participants]
  Never | 63
  Quit | 43
  Currently Use | 19
  Missing | 0

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) Change From Baseline
Description: Evaluation of the change of the Back VAS, Hip VAS and the Leg VAS at the 24 month post-operative visit as compared to pre-op time periods. Information on all reports of pain/numbness/tingling and the location of symptoms were captured and evaluated.
  VAS scale ranged from 0 - 10cm with the 10cm accounting for the highest level of pain.
Time Frame: 24 months
Population: All patients were accounted for
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Back: Evaluation of the improvement of the Back VAS at the 24 month post-operative visit as compared to pre-op time periods. Information on all reports of pain/numbness/tingling and the location of symptoms was captured and evaluated.
- Left Hip: Evaluation of the improvement of the Left Hip VAS at the 24 month post-operative visit as compared to pre-op time periods. Information on all reports of pain/numbness/tingling and the location of symptoms was captured and evaluated.
- Right Hip: Evaluation of the improvement of the Right Hip VAS at the 24 month post-operative visit as compared to pre-op time periods. Information on all reports of pain/numbness/tingling and the location of symptoms was captured and evaluated.
- Left Leg: Evaluation of the improvement of the Left Leg VAS at the 24 month post-operative visit as compared to pre-op time periods. Information on all reports of pain/numbness/tingling and the location of symptoms was captured and evaluated.
- Right Leg: Evaluation of the improvement of the Right Leg VAS at the 24 month post-operative visit as compared to pre-op time periods. Information on all reports of pain/numbness/tingling and the location of symptoms was captured and evaluated.
Arm/Group | Back | Left Hip | Right Hip | Left Leg | Right Leg
Number analyzed (Participants) | 56 | 56 | 56 | 56 | 56
score on a scale | -4.3 (3.7) | -2.3 (3.8) | -4.0 (3.7) | -2.1 (3.4) | -3.5 (4)

2. Primary Outcome: Number of Patients With Adverse Events AEs)
Description: The evaluation of all adverse events including device related, procedure related and additional serious adverse events.
Time Frame: Operative to 24 month
Population: This is an analysis of the number of participants that reported any form of adverse event. Participants were evaluated for all adverse events including device related, procedure related, and additional serious adverse events.
  9 of the 30 SAE participants did not experience a non-SAE events. The other 21 participants had events in both categories
Measure: Number; unit: participants
Groups:
- Up to Post-Operative: Number of Patients with Adverse Events up to Post-Operative
- Post-Operative to 3 Months: Number of Patients with Adverse Events Post-Operative to 3 Months
- 3 to 6 Months: Number of Patients with Adverse Events 3 to 6 Months
- 6 to 12 Months: Number of Patients with Adverse Events 6 to 12 Months
- 12 to 24+ Months: Number of Patients with Adverse Events 12 to 24+ Months
- Overall: Overall number of Patients with Adverse Events
Arm/Group | Up to Post-Operative | Post-Operative to 3 Months | 3 to 6 Months | 6 to 12 Months | 12 to 24+ Months | Overall
Number analyzed (Participants) | 125 | 125 | 125 | 125 | 125 | 125
participants
  Any AE | 45 | 16 | 22 | 33 | 23 | 82
  Any AE : Procedure Related | 23 | 3 | 4 | 6 | 4 | 34
  Any AE : Device Related | 4 | 2 | 3 | 2 | 2 | 10
  Any AE : Mild | 28 | 7 | 7 | 19 | 9 | 51
  Any AE : Moderate | 21 | 7 | 15 | 12 | 14 | 52
  Any AE : Severe | 5 | 4 | 3 | 5 | 6 | 20
  Any Serious Adverse Event (SAE) | 10 | 4 | 3 | 7 | 10 | 30
  Any SAE : Procedure Related | 4 | 0 | 0 | 1 | 1 | 6
  Any SAE : Device Related | 1 | 1 | 0 | 0 | 1 | 2
  Any SAE : Mild | 3 | 0 | 0 | 1 | 2 | 6
  Any SAE : Moderate | 4 | 1 | 1 | 1 | 3 | 10
  Any SAE : Severe | 5 | 3 | 2 | 5 | 6 | 18

3. Secondary Outcome: Change in Pain/Dysesthesia Score From Baseline (Pre-Operative)
Description: Neurological evaluation of the patient, with specific evaluation of psoas muscle weakness, radiating radicular pain, knee extension weakness, dorsiflexion weakness, plantarflexion weakness and anterior thigh numbness was performed using Patient symptom Questionnaire (0-100mm analog scale with 100mm being the highest pain/weakness/numbness)
Time Frame: time of discharge, an average of 4.5 days, up to 8 weeks post-operatively, 3 months, 6 months, 12 months, 24 months
Population: The overall number of patients participated in each interval differed from the number of patients that were evaluated for the body location measurements.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Discharge; Post-Operative; 3 Months; 6 Months; 12 Months; 24 Months: Neurological evaluation of the patient, with specific evaluation of psoas muscle weakness, radiating radicular pain, knee extension weakness, dorsiflexion weakness, plantarflexion weakness and anterior thigh numbness
Arm/Group | Discharge | Post-Operative | 3 Months | 6 Months | 12 Months | 24 Months
Number analyzed (Participants) | 92 | 117 | 107 | 103 | 93 | 56
score on a scale
  Pain Above Left Knee: number analyzed (Participants) | 88 | 111 | 103 | 98 | 90 | 54
  Pain Above Left Knee | -3.9 (28.6) | -14.3 (38.2) | -20 (34.3) | -18.7 (33.8) | -22.4 (34.6) | -17.8 (34)
  Pain Above Right Knee: number analyzed (Participants) | 88 | 112 | 104 | 99 | 91 | 54
  Pain Above Right Knee | -15.3 (33.8) | -21.3 (35.8) | -26.9 (33.9) | -29.2 (33.9) | -31 (31.4) | -31.2 (31.8)
  Left Groin Pain: number analyzed (Participants) | 87 | 108 | 102 | 97 | 89 | 53
  Left Groin Pain | -0.3 (28.3) | -10.4 (33.5) | -11.8 (30.8) | -14.5 (28.7) | -15.1 (31.1) | -10.8 (25.2)
  Right Groin Pain: number analyzed (Participants) | 86 | 109 | 102 | 97 | 90 | 54
  Right Groin Pain | -7.2 (29.9) | -15.1 (33.4) | -15.7 (31.6) | -19.9 (33.1) | -20.3 (31) | -23.2 (30.5)
  Flexing Left Hip Weakness | 7.8 (37.9) | -10.6 (39.7) | -15.1 (33.3) | -17.8 (33.2) | -20.0 (32.2) | -12.5 (29.2)
  Flexing Right Hip Weakness | -0.3 (34.1) | -17.3 (34.7) | -17.6 (34.0) | -23.5 (33.8) | -24.7 (31.7) | -20.4 (34.1)
  Extending Left Hip Weakness | 8.6 (39.7) | -7.4 (40.1) | -14.0 (30.1) | -16.9 (30.7) | -16.8 (33.4) | -11.0 (30.6)
  Extending Right Hip Weakness | -2.8 (33.1) | -15.6 (36.2) | -16.2 (36.5) | -24.4 (32.3) | -24.4 (33.1) | -22.4 (34.9)
  Left Hip Stairs Weakness: number analyzed (Participants) | 86 | 117 | 107 | 102 | 92 | 56
  Left Hip Stairs Weakness | 6.1 (38) | -15.9 (42.5) | -20.5 (38.9) | -24.7 (36.8) | -26.8 (36.6) | -20.0 (33.7)
  Right Hip Stairs Weakness: number analyzed (Participants) | 86 | 117 | 107 | 102 | 92 | 56
  Right Hip Stairs Weakness | 0.4 (36.2) | -20.7 (39.6) | -24.3 (37.7) | -29.7 (36.4) | -30.1 (35.2) | -27.8 (35.5)
  Left Hip Cross Leg Weakness: number analyzed (Participants) | 89 | 116 | 107 | 103 | 92 | 56
  Left Hip Cross Leg Weakness | 16.8 (41.1) | -8.2 (42.7) | -16.7 (40.1) | -21.0 (34.7) | -25.5 (36.3) | -19.2 (31.8)
  Right Hip Cross Leg Weakness: number analyzed (Participants) | 89 | 116 | 107 | 103 | 92 | 56
  Right Hip Cross Leg Weakness | 6.1 (37.1) | -13.4 (39.0) | -21.6 (36.5) | -25.2 (35.8) | -27.8 (32.4) | -25.6 (32.8)

4. Secondary Outcome: Change in Oswestry Disability Index From Baseline (Pre-Operative)
Description: The Oswestry Disability Index (ODI) is a validated instrument including items that relate to subjective symptomatology and activities of daily living (pain intensity, personal care, lifting, walking, sitting, standing, sex life, traveling). This patient-reported outcome measure is a 10 item questionnaire that evaluates disability and functional impairment associated with back problems. Each item is scored from O up to 5, with higher scores corresponding to greater disability. A total ODI score is determined by adding the scores of the individual questions and dividing that total by the maximum possible score (i.e., 50 if all questions are answered) to yield a percentage. Therefore, the ODI score ranges from 0% to 100%.
Time Frame: time of discharge, an average of 4.5 days, up to 8 weeks post-operatively, 3 months, 6 months, 12 months, 24 months
Population: 131 patients started the study at Pre-op, 6 patients did not complete the survey; 125 started operative, 34 patients did not complete the survey at Discharge; 121 started the Post-operative interval, 4 patients did not complete the survey; 111 patients started at 3 Month interval, 4 patients did not complete the survey; All patients who started at 6 months and 24 months completed their surveys at their respective intervals.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Discharge; Post-Operative; 3 Months; 6 Months; 12 Months; 24 Months: Change in Oswestry Disability Index
Arm/Group | Discharge | Post-Operative | 3 Months | 6 Months | 12 Months | 24 Months
Number analyzed (Participants) | 91 | 117 | 107 | 104 | 93 | 56
score on a scale | 7.7 (19.5) | -10.1 (21.1) | -17.3 (18.5) | -22.7 (19) | -26.9 (17.5) | -24.3 (17.6)

5. Secondary Outcome: Change in Health-Related Quality of Life From Baseline (Pre-op)
Description: Health-related quality of life was evaluated in all study subjects using the SF-12v2 Health Survey. This shortened and simplified version of the SF-36 makes the questionnaire less ambiguous for patients. It has a self-administered form that makes it easy to read and complete, and that reduces missing responses. The physical and mental component summary scales, referred to as PCS-12 and MCS-12 were evaluated against published normative values and a 15% improvement in these scores was used as an assessment of success. In calculating the true value of a treatment, the scores from the SF-12v2 were converted into a utility index (SF-6D), which considered not only how many years a medical intervention could have added to a patient's life, but also the quality of that life. Use of the SF-6D did not expand the questions administered to the patients. The scale ranged from 0-100% with 100% being the best quality of life.
Time Frame: time of discharge, an average of 4.5 days, up to 8 weeks post-operatively, 3 months, 6 months, 12 months, 24 months
Population: The number analyzed in Mental Health and Physical Health rows for 6 Months and 12 Months differ due to the inability for a participant to complete the required forms for those two intervals.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Discharge; Post-Operative; 3 Months; 6 Months; 12 Months; 24 Months: Change in Health-Related Quality of Life From Baseline
Arm/Group | Discharge | Post-Operative | 3 Months | 6 Months | 12 Months | 24 Months
Number analyzed (Participants) | 91 | 117 | 106 | 104 | 92 | 56
score on a scale
  Mental Health | 0.01 (10) | 4.0 (12.4) | 4.8 (11.6) | 7.6 (12.7) | 7.6 (10.7) | 7.1 (11.9)
  Physical Health: number analyzed (Participants) | 91 | 117 | 106 | 103 | 91 | 56
  Physical Health | 0.6 (6.8) | 4.6 (9.3) | 8.2 (9.2) | 9.7 (11.5) | 12.9 (9) | 11.5 (10.1)

6. Secondary Outcome: Radiographic Assessments
Description: Quantitative and qualitative radiographic assessment of the pre and post-operative AP, and Lateral, Flexion/Extension images were performed. Radiographic and qualitative assessments performed include:
  * Device Condition: looks at both the cage inside the vertebrae and the hardware outside the vertebrae. It looks at whether or not the device is intact or not (subsidence or migration)
  * Fusion/Non-fusion: whether bone has grown within the space between the spinal vertebrae. If fusion occurs, it results in Bony Bridging
Time Frame: 12 mo to 24 mo
Population: The numbers are different from the overall number analyzed due to the different number of people who participated in each visit's radiographic analysis
Measure: Count of Participants; unit: Participants
Groups:
- Level 1: One vertebrae level analyzed
- Superior: Analysis of the upper level of a two-level vertebrae
- Inferior: Analysis of the lower level of a two-level vertebrae
Arm/Group | Level 1 | Superior | Inferior
Number analyzed (Participants) | 95 | 23 | 23
Participants
  12 Month Fusion: number analyzed (Participants) | 60 | 18 | 18
  12 Month Fusion: Absent | 2 | 3 | 3
  12 Month Fusion: Partial Consolidation | 10 | 2 | 2
  12 Month Fusion: Bridging / Fusion | 33 | 11 | 11
  12 Month Fusion: Intact | 0 | 0 | 0
  12 Month Fusion: Loosening | 0 | 0 | 0
  12 Month Fusion: Fracture | 0 | 0 | 0
  12 Month Fusion: Not Applicable | 0 | 0 | 0
  12 Month Fusion: Unable to Assess | 15 | 2 | 2
  12 Month Fusion: Subsidence | 0 | 0 | 0
  12 Month Fusion: Migration | 0 | 0 | 0
  12 Month Fusion: Subsidence & Migration | 0 | 0 | 0
  12 Month Fusion: Other | 0 | 0 | 0
  24 Month Fusion: number analyzed (Participants) | 31 | 13 | 13
  24 Month Fusion: Absent | 0 | 1 | 1
  24 Month Fusion: Partial Consolidation | 0 | 0 | 0
  24 Month Fusion: Bridging / Fusion | 29 | 12 | 12
  24 Month Fusion: Intact | 0 | 0 | 0
  24 Month Fusion: Loosening | 0 | 0 | 0
  24 Month Fusion: Fracture | 0 | 0 | 0
  24 Month Fusion: Not Applicable | 0 | 0 | 0
  24 Month Fusion: Unable to Assess | 0 | 0 | 0
  24 Month Fusion: Subsidence | 2 | 0 | 0
  24 Month Fusion: Migration | 0 | 0 | 0
  24 Month Fusion: Subsidence & Migration | 0 | 0 | 0
  24 Month Fusion: Other | 0 | 0 | 0
  12 Month Hardware Condition: number analyzed (Participants) | 60 | 18 | 18
  12 Month Hardware Condition: Absent | 0 | 0 | 0
  12 Month Hardware Condition: Partial Consolidation | 0 | 0 | 0
  12 Month Hardware Condition: Bridging / Fusion | 0 | 0 | 0
  12 Month Hardware Condition: Intact | 48 | 17 | 17
  12 Month Hardware Condition: Loosening | 0 | 1 | 1
  12 Month Hardware Condition: Fracture | 0 | 0 | 0
  12 Month Hardware Condition: Not Applicable | 11 | 0 | 0
  12 Month Hardware Condition: Unable to Assess | 1 | 0 | 0
  12 Month Hardware Condition: Subsidence | 0 | 0 | 0
  12 Month Hardware Condition: Migration | 0 | 0 | 0
  12 Month Hardware Condition: Subsidence & Migration | 0 | 0 | 0
  12 Month Hardware Condition: Other | 0 | 0 | 0
  24 Month Hardware Condition: number analyzed (Participants) | 31 | 13 | 13
  24 Month Hardware Condition: Absent | 0 | 0 | 0
  24 Month Hardware Condition: Partial Consolidation | 0 | 0 | 0
  24 Month Hardware Condition: Bridging / Fusion | 0 | 0 | 0
  24 Month Hardware Condition: Intact | 28 | 12 | 12
  24 Month Hardware Condition: Loosening | 0 | 1 | 1
  24 Month Hardware Condition: Fracture | 0 | 0 | 0
  24 Month Hardware Condition: Not Applicable | 3 | 0 | 0
  24 Month Hardware Condition: Unable to Assess | 0 | 0 | 0
  24 Month Hardware Condition: Subsidence | 0 | 0 | 0
  24 Month Hardware Condition: Migration | 0 | 0 | 0
  24 Month Hardware Condition: Subsidence & Migration | 0 | 0 | 0
  24 Month Hardware Condition: Other | 0 | 0 | 0
  12 Month Cage Condition: number analyzed (Participants) | 60 | 18 | 18
  12 Month Cage Condition: Absent | 0 | 0 | 0
  12 Month Cage Condition: Partial Consolidation | 0 | 0 | 0
  12 Month Cage Condition: Bridging / Fusion | 0 | 0 | 0
  12 Month Cage Condition: Intact | 58 | 16 | 15
  12 Month Cage Condition: Loosening | 0 | 0 | 0
  12 Month Cage Condition: Fracture | 0 | 0 | 0
  12 Month Cage Condition: Not Applicable | 0 | 0 | 0
  12 Month Cage Condition: Unable to Assess | 0 | 0 | 0
  12 Month Cage Condition: Subsidence | 2 | 1 | 1
  12 Month Cage Condition: Migration | 0 | 0 | 1
  12 Month Cage Condition: Subsidence & Migration | 0 | 1 | 0
  12 Month Cage Condition: Other | 0 | 0 | 1
  24 Month Cage Condition: number analyzed (Participants) | 31 | 13 | 13
  24 Month Cage Condition: Absent | 0 | 0 | 0
  24 Month Cage Condition: Partial Consolidation | 0 | 0 | 0
  24 Month Cage Condition: Bridging / Fusion | 0 | 0 | 0
  24 Month Cage Condition: Intact | 31 | 13 | 11
  24 Month Cage Condition: Loosening | 0 | 0 | 0
  24 Month Cage Condition: Fracture | 0 | 0 | 0
  24 Month Cage Condition: Not Applicable | 0 | 0 | 0
  24 Month Cage Condition: Unable to Assess | 0 | 0 | 0
  24 Month Cage Condition: Subsidence | 0 | 0 | 1
  24 Month Cage Condition: Migration | 0 | 0 | 0
  24 Month Cage Condition: Subsidence & Migration | 0 | 0 | 0
  24 Month Cage Condition: Other | 0 | 0 | 1

7. Secondary Outcome: Patient Satisfaction
Description: At the 12 month and 24 month follow-up visits, subjects were asked whether they were satisfied with the outcome of their surgery (Yes/No) and whether they would repeat the operation (Yes/No).
Time Frame: 12 month and 24 month
Population: Patient self-assessment of the procedure at 12M and 24M
Measure: Count of Participants; unit: Participants
Groups:
- 12 Month: Patient satisfaction at 12 Month
- Repeat Procedure: Patient satisfaction at 24 Month
Arm/Group | 12 Month | Repeat Procedure
Number analyzed (Participants) | 97 | 56
Participants
  Satisfied: Yes | 80 | 51
  Satisfied: No | 11 | 5
  Satisfied: Not Reported | 6 | 0
  Repeat Procedure: Yes | 80 | 51
  Repeat Procedure: No | 11 | 5
  Repeat Procedure: Not Reported | 6 | 0

8. Secondary Outcome: Odom's Criteria
Description: At the 24 month follow-up visit, the Investigator rated the clinical disposition of each study subject according to Odom's Criteria as follows:
  Excellent: all pre-operative symptoms relieved, able to carry out daily occupations without impairment.
  Good: minimum persistence of pre-operative symptoms, able to carry out daily occupations without significant interference.
  Fair/Satisfactory: relief of some pre-operative symptoms but physical activity is significantly limited.
  Poor: symptoms or signs unchanged or worse.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Groups:
- 24 Month: Odom's criteria
Arm/Group | 24 Month
Number analyzed (Participants) | 56
Participants
  Excellent | 33
  Good | 17
  Fair/Satisfactory | 5
  Not Reported | 1

9. Secondary Outcome: Surgery Time
Description: The length of the surgical procedure from the initial incision to final closure were captured from the Anesthesia Record.
Time Frame: During operation.
Population: 3 of 125 subjects did not have surgery time included. There were 12 staged procedures increasing the overall number of procedures to 134
Measure: Mean (Standard Deviation); unit: Minutes
Units Other Than Participants: surgeries
Groups:
- Surgery Time: The length of the surgical procedure
Arm/Group | Surgery Time
Number analyzed (Participants) | 122
Number analyzed (surgeries) | 134
Minutes | 142 (62.7)

10. Secondary Outcome: Anesthesia Time
Description: The length of time the patient is under anesthesia were captured from the Anesthesia Record.
Time Frame: During operation.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Minutes
Units Other Than Participants: surgeries
Groups:
- Anesthesia Time: The length of time the patient is under anesthesia
Arm/Group | Anesthesia Time
Number analyzed (Participants) | 122
Number analyzed (surgeries) | 134
Minutes | 219.8 (84.9)

11. Secondary Outcome: Estimated Blood Loss
Description: The amount of blood loss over the entire length of the surgery, documented on the Anesthesia Record, was captured.
Time Frame: During Operation
Population: 11 of 125 subjects did not have blood loss included. There were 12 staged procedures increasing the overall number of procedures to 126.
Measure: Mean (Standard Deviation); unit: Cubic Centimeters
Units Other Than Participants: surgeries
Groups:
- Estimated Blood Loss: The amount of blood loss over the entire length of the surgery
Arm/Group | Estimated Blood Loss
Number analyzed (Participants) | 114
Number analyzed (surgeries) | 126
Cubic Centimeters | 76.5 (78.9)

12. Secondary Outcome: Number of Participants With Abnormal Neuromonitoring System Results
Description: Abnormal result(s) of neuromonitoring systems (Train of Four, Electromyography (EMG), Triggered EMG, Somato Sensory Evoked Potential (SSEP) and Motor Evoked Potential (MEP)) utilized during the surgery were captured.
Time Frame: During operation
Measure: Count of Participants; unit: Participants
Groups:
- Train of Four; Electromyography (EMG); Triggered EMG; Somato Sensory Evoked Potential (SSEP); Motor Evoked Potential (MEP): Abnormal result(s) of neuromonitoring systems utilized during the surgery
Arm/Group | Train of Four | Electromyography (EMG) | Triggered EMG | Somato Sensory Evoked Potential (SSEP) | Motor Evoked Potential (MEP)
Number analyzed (Participants) | 85 | 121 | 119 | 75 | 30
Participants | 1 | 0 | 0 | 0 | 0

13. Secondary Outcome: Length of Hospital Stay
Description: The length of hospital stay from the date of hospital admission to the date of discharge was calculated.
Time Frame: From admission to discharge
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Length of Hospital Stay: The length of hospital stay from the date of hospital admission to the date of discharge
Arm/Group | Length of Hospital Stay
Number analyzed (Participants) | 125
Days | 4.5 (3.3)

14. Secondary Outcome: Change in Work/School Status Compared to Baseline
Description: The ability to and the time it takes for the subject to be cleared to return to work/school from the date of surgery was documented.
Time Frame: Pre-operative to 24 months
Population: All patients who participated in each interval were accounted for including the missing category
Measure: Count of Participants; unit: Participants
Groups:
- Pre-Op; Initial Post-Operative; 3 Months; 6 Months; 12 Months; 24 Months: The ability to and the time it takes for the subject to be cleared to return to work/school from the date of surgery
Arm/Group | Pre-Op | Initial Post-Operative | 3 Months | 6 Months | 12 Months | 24 Months
Number analyzed (Participants) | 125 | 122 | 111 | 104 | 97 | 56
Participants
  Unemployed, unrelated to back/leg conditions | 16 | 25 | 22 | 22 | 16 | 8
  Not attending work/school by choice | 42 | 35 | 36 | 31 | 35 | 21
  Unable to go due to back/leg pain/conditions | 30 | 41 | 24 | 18 | 16 | 10
  Attending work/school with some restrictions | 25 | 15 | 14 | 15 | 8 | 5
  Attending work/school with no restrictions | 12 | 5 | 14 | 17 | 20 | 12
  Missing | 0 | 1 | 1 | 1 | 2 | 0

15. Secondary Outcome: Change in Use of Narcotics Post-Surgery Compared to Baseline
Description: The types and dosages of any narcotics taken by the patient post-surgery were documented.
Time Frame: Pre-operative to 24 months
Population: All patients who participated in each interval were accounted for including the missing category
Measure: Count of Participants; unit: Participants
Groups:
- Pre-Op; Initial Post-Operative; 3 Months; 6 Months; 12 Months; 24 Months: The types and dosages of any narcotics taken by the patient post-surgery
Arm/Group | Pre-Op | Initial Post-Operative | 3 Months | 6 Months | 12 Months | 24 Months
Number analyzed (Participants) | 125 | 122 | 111 | 104 | 97 | 56
Participants
  Back Meds: None | 15 | 15 | 23 | 26 | 30 | 24
  Back Meds: Non-narcotics or NSAIDs | 42 | 20 | 25 | 28 | 29 | 14
  Back Meds: Intermittent short-acting narcotics | 21 | 38 | 34 | 27 | 16 | 7
  Back Meds: Chronic daily short-acting narcotics | 30 | 24 | 20 | 17 | 15 | 9
  Back Meds: Chronic daily long-acting narcotics | 16 | 19 | 7 | 6 | 3 | 1
  Back Meds: IV or injected narcotics | 1 | 6 | 1 | 0 | 1 | 1
  Back Meds: Missing | 0 | 0 | 1 | 0 | 3 | 0
  Non-Back Meds: None | 103 | 97 | 90 | 79 | 64 | 41
  Non-Back Meds: Non-narcotics or NSAIDs | 14 | 14 | 11 | 17 | 22 | 12
  Non-Back Meds: Intermittent short-acting narcotics | 2 | 4 | 6 | 5 | 7 | 1
  Non-Back Meds: Chronic daily short-acting narcotics | 5 | 5 | 2 | 2 | 1 | 2
  Non-Back Meds: Chronic daily long-acting narcotics | 1 | 2 | 0 | 1 | 0 | 0
  Non-Back Meds: IV or injected narcotics | 0 | 0 | 1 | 0 | 0 | 0
  Non-Back Meds: Missing | 0 | 0 | 1 | 0 | 3 | 0

ADVERSE EVENTS:
Time Frame: Operative to 24+ Months
Description: Any untoward medical occurrence in a subject undergoing surgery in this trial which does not necessarily have a causal relationship with this intervention. An AE can, therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the one of the devices. Any AE that occurs during the subject's participation in the study will be recorded on the Adverse Event case report form.
Groups:
- Participants With Adverse Events: Participants were evaluated for all adverse events including device related, procedure related, and additional serious adverse events.
  9 of the 30 SAE participants did not experience a non-SAE events. The other 21 participants had events in both categories.
  The study did not establish a frequency threshold, therefore, all AEs are listed.
Arm/Group | Participants With Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/125
Serious Adverse Events (participants affected / at risk) | 30/125
Other Adverse Events (participants affected / at risk) | 73/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Adverse Events (N=125)
Cardiac failure (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Adjacent segment degeneration (Injury, poisoning and procedural complications) | 1 (1)
Cerebrospinal fluid leakage (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (6)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Cervical cord compression (Nervous system disorders) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 1 (1)
Dural tear (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1)
Lumbar spinal stenosis (Nervous system disorders) | 2 (2)
Metabolic encephalopathy (Nervous system disorders) | 1 (2)
Syncope (Nervous system disorders) | 1 (1)
Device dislocation (Product Issues) | 2 (3)
Confusional state (Psychiatric disorders) | 1 (1)
Bladder dysfunction (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Wound drainage (Surgical and medical procedures) | 2 (2)
Carpal tunnel decompression (Surgical and medical procedures) | 1 (2)
Cholecystectomy (Surgical and medical procedures) | 1 (1)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1)
Medical device removal (Surgical and medical procedures) | 2 (2)
Pituitary tumour removal (Surgical and medical procedures) | 1 (1)
Spinal decompression (Surgical and medical procedures) | 1 (1)
Spinal fusion surgery (Surgical and medical procedures) | 2 (2)
Spinal laminectomy (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Adverse Events (N=125)
Anaemia postoperative (Blood and lymphatic system disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Eyelid ptosis (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anorectal disorder (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Discomfort (General disorders) | 1 (2)
Dysplasia (General disorders) | 1 (1)
Fat necrosis (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Nodule (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 4 (4)
Swelling (General disorders) | 1 (1)
Tissue injury (General disorders) | 2 (4)
Hepatic lesion (Hepatobiliary disorders) | 1 (1)
Abscess (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5)
Wound infection (Infections and infestations) | 3 (3)
Eye contusion (Injury, poisoning and procedural complications) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 11 (13)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accidents (Injury, poisoning and procedural complications) | 1 (1)
skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Osteoporosis (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (16)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (25)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 (2)
Meniscus injury (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle injury (Musculoskeletal and connective tissue disorders) | 2 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13 (16)
Neck pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (24)
Pseuarthrosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Spinal compression fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 1 (1)
Dural tear (Nervous system disorders) | 1 (1)
Dysaesthesia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 7 (8)
Lumbar radiculopathy (Nervous system disorders) | 1 (1)
Lumbar spinal stenosis (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (2)
Paraesthesia (Nervous system disorders) | 2 (2)
Peroneal nerve palsy (Nervous system disorders) | 2 (3)
Piriformis syndrome (Nervous system disorders) | 1 (1)
Spinal claudication (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Vertebral foraminal stenosis (Nervous system disorders) | 1 (1)
Device failure (Product Issues) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Attention deficit / hyperactivity disorder (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Obsessive-compulsive disorder (Psychiatric disorders) | 1 (1)
Bladder dysfunction (Renal and urinary disorders) | 1 (2)
Urinary retention (Renal and urinary disorders) | 4 (5)
Orchitis (Reproductive system and breast disorders) | 1 (1)
Testicular swelling (Reproductive system and breast disorders) | 1 (1)
Uterine leiomyoma (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Blepharoplasty (Surgical and medical procedures) | 1 (1)
Corneal suture (Surgical and medical procedures) | 1 (1)
Incisional drainage (Surgical and medical procedures) | 1 (1)
Spinal fusion (Surgical and medical procedures) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Ecchymosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Haemorrhoidal haemorrhage (Vascular disorders) | 1 (1)
Rectal haemorrhage (Vascular disorders) | 1 (1)
Uterine haemorrhage (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution/PI shall not disclose/use any confidential/proprietary information (CI) disclosed to/developed by the Institution during the study. Institution/PI agree to hold the results of the Study in confidence, and shall not disclose them except with prior written consent of K2M. Institution agrees to submit any Articles to K2M for review prior to publication and agrees to edit out any confidential information identified by K2M.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-27): https://cdn.clinicaltrials.gov/large-docs/29/NCT02068729/Prot_SAP_000.pdf